CLINICAL TRIAL: NCT00422357
Title: Effect of Urtica Dioica on Glycemic Control in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NNFTRI-1385
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Urtica Dioica (or stinging nettle); Hypoglycemic agents
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Urtica Dioica (Tea bag)

SUMMARY:
Diabetes mellitus is the most common metabolic disorder worldwide. Some herbs are traditionally used in treatment of type 2 diabetes mellitus (T2DM). Urtica Dioica (UD) or stinging nettle is traditionally used in Morocco, Turkey, Brasil, Jordan and with much frequency in northern Iran.

Studies on animal models along with in vitro studies has shown hypoglycemic effect for aqueous extract of UD.

This study aimed to investigate hypoglycemic effects of UD tea bags in patients with T2DM on glycemic control, insulin sensitivity, along with its effects on lipid profile (LP), blood pressure (BP), liver, and kidney function.

DETAILED DESCRIPTION:
The study will be performed under randomized, double-blind, placebo controlled, and case-control design. The object of this study is patients with T2DM. Patients are randomly assigned to start with placebo tea bags (3 tea bags as 2-gram tea bag steamed in boiling water for 20 minutes: mixture of bran powder which is already boiled in water twice plus spinach powder) in control groups and UD tea bags (3 tea bags as 2-gram tea bag steamed in boiling water for 20 minutes) in patients with T2DM for two months. Every two weeks, fasting glucose, postprandial glucose after a standard breakfast, serum insulin, lipids, alanine amino transferase (ALT), aspartate amino transferase (AST), creatinine (to calculate GFR), along with blood pressure will be measured.

To the best of our knowledge, this is the first Randomized Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM
* Must be able to drink UD or Placebo tea bags 3 times every day

Exclusion Criteria:

* Insulin dependent diabetes
* History of congestive heart failure within last 5 years (NYHA Class III-IV)
* History of significant pulmonary disease, myocardial infarction, cerebrovascular accident, or nephrotic syndrome within last 1 year
* Thyroid disease
* Known renal or hepatic insufficiency
* Gastric problem
* History of UD or and other herb use in past 6 months
* Pregnancy or lactation
* Use of any herbal or supplement within past 6 months
* Use of an investigational drug (within 30 days prior to enrollment)
* Known maternal allergies
* Dumping syndrome

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2007-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose every two weeks.
Post prandial blood glucose every two weeks.
Fasting insulin every two weeks.
Insulin sensitivity as Quantitative Insulin Sensitivity Check Index (QUIKI) every two weeks.
C-Peptide every two weeks.
HBA1C every two weeks.
Serum lipids every two weeks.
Liver enzymes (ALT, AST) every two weeks.
GFR every two weeks.
Blood pressure every two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Rastmanesh, Ph.D., Study Chair — Shahid Beheshti University of Medical Sciences; Navid Saadat, MD, Study Director — Shaheed Beheshti Medical Univrsity
Locations (1):
- Primary Health Care Office, Mahmood-Abaad, Mazandaran, Iran